CLINICAL TRIAL: NCT00978237
Title: CT to Assess the Effect on the Subcutaneous Fat of Change of EFV for LPV/r in HIV-infected Patients Who Developed Lipoatrophy and Remains Despite Treatment With Efavirenz and Fixed-dose Combination of no Thymidine Nucleoside Analogues.
Brief Title: Clinical Trial to Assess the Effect of the Change of Efavirenz (EFV) for Lopinavir/Ritonavir (LPV/r) in Lipoatrophy in HIV-infected Patients
Acronym: LIPOKAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIPOKAL
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections; Lipoatrophy
Keywords: HIV - Lipoatrophy; treatment experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFV and Fixed combinations of analogues (Active Comparator): EFV + Fixed combinations of analogue tenofovir + emtricitabine, or abacavir + lamivudine
  Interventions: Drug: EFV
- LPV/r and combination of analogues. (Experimental)
  Interventions: Drug: LPV/r

INTERVENTIONS:
Drug: EFV — one pill QD VO.
  Arms: EFV and Fixed combinations of analogues
Drug: LPV/r — 2 pills QD VO
  Arms: LPV/r and combination of analogues.

SUMMARY:
Eligible HIV-infected patients with clinically evident lipoatrophy despite treatment with efavirenz and fixed-dose combination of thymidine nucleoside analogues will be informed and asked to enroll in the study; will be randomized (1:1) into two branches, A: EFV + Fixed combinations of analogue tenofovir + emtricitabine.B (experimental): LPV/r + combination of correspondent analogues. The main variable is the evaluation of the absolute change in limb fat mass at 24 months from baseline in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients HIV positive > 18 years.
* Patients in treatment with Sustiva(r)+Truvada(r); or Sustiva (r)+Kivexa(r).
* HIV-ARN < 50 copies/mL in the las six months.
* Clinically evident lipoatrophy (moderate or severe).
* Negative pregnancy test.
* Signed informed consent.

Exclusion Criteria:

* Evidence of failure or mutation to therapy with protease inhibitors.
* Patients that can not be treated with LPV/r.
* Mild lipoatrophy.
* History of alcoholism or drug addiction that discourages participation in the study.
* Pregnancy or breastfeeding.
* Documented current or 4 weeks prior opportunistic infection.
* Creatinin clearance < 60mL/min.
* Concomitant use of nephrotoxic drugs or immunosuppressants.
* Actual treatment with systemic corticosteroids, IL-2 or chemotherapy.
* Patients under treatment with other drugs in investigation.
* Acute hepatitis.
* Any other disease that discourages participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Absolute change in limb fat mass measured by DEXA. | 24 months.

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Central de Asturias, Asturias
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Fe, Valencia
  - Hospital Xeral-Cíes, Vigo

REFERENCES:
- [Derived] Rojas J, Lonca M, Imaz A, Estrada V, Asensi V, Miralles C, Domingo P, Montero M, del Rio L, Fontdevila J, Perez I, Cruceta A, Gatell JM, Arnedo M, Martinez E. Improvement of lipoatrophy by switching from efavirenz to lopinavir/ritonavir. HIV Med. 2016 May;17(5):340-9. doi: 10.1111/hiv.12314. Epub 2015 Sep 10. PMID 27089862